CLINICAL TRIAL: NCT06698848
Title: Integrating Ketamine Effects on Neuronal Molecular Signatures and the Brain Functional and Structural Connectome
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Amit Anand, BWPO Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P001580
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Depression; Suicide
MeSH Terms: conditions — Depression; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous Ketamine (Experimental): Intravenous ketamine will be given at a dose of 0.5 mg/kg over 40 minutes with a maximum dose of 60 mg.
  Interventions: Drug: ketamin

INTERVENTIONS:
Drug: ketamin — Participants in this study will have been diagnosed with major depressive episode (MDE) and have not received any psychiatric treatment for at least 2 weeks (5 weeks if on fluoxetine).Patients will receive intravenous ketamine as the only study drug treatment for the 2 weeks of the study. Magnetic Resonance Imaging (MRI) will be used to measure effects of ketamine on brain structure, function and chemistry, in addition to a soft-nasal brushing procedure to obtain olfactory sensory neurons which will provide the ability to profile in vivo how neurons may react to KET treatment in depressed patients.

SUMMARY:
Subanesthetic dose of intravenous ketamine (KET) has been found to be highly effective in rapid treatment depression and associated suicidality but its exact mechanism of remains uncertain. This study will use a novel approach to elucidate KET's effects on the molecular/ gene expression pathways in living neurons obtained from the olfactory epithelium and correlate the changes to rapid improvement in depression via changes in the brain connectome. The study will identify the molecular targets and pathways involved in KET'S mechanism of rapid clinical action and pave the way for development of novel, more efficacious, and safer therapeutic agents.

DETAILED DESCRIPTION:
We propose a mechanistic clinical trial to identify molecular and imaging correlates of rapid action of intravenous subanesthetic dose of ketamine (KET). KET is a rapidly acting highly effective treatment for depression and frequently accompanying suicidality. However, its mechanism of rapid action remains unclear which has hindered development of methods to monitor its effects and development of new medications with similar efficacy but more favorable side-effects profile. A basic science bottom-up approach for identification and development of novel drug agents has a high degree of uncertainty. Therefore, a reverse translational approach that first identifies drug targets in humans holds promise. Our clinical translational program has developed a method to integrate drug related molecular, brain imaging and clinical changes in patients to identify novel drug targets for psychiatric illnesses. We have successfully used this method in vivo to characterize mechanism of action of lithium - a gold standard drug for bipolar disorder. In this application, we propose to apply the method to KET's mechanism of rapid action in the treatment of depression. Clinical efficacy of KET in depression and its complex effects on multiple brain physiological functions may be best deciphered using a network properties-metric approach. This approach is critical because it provides insight into the function of complex brain networks (e.g., graph theory metrics provide summary measures of whole-brain and local network properties), which is more likely to be closely linked to complex brain behavioral states such as depression. Furthermore, the relationship between neuroimaging effects of ketamine and its molecular effects in humans has been even less studied. This proposal addresses these important gaps in knowledge. We will study 90 depressed subjects (medication-free for 2 weeks) at baseline and after 3 alternate-day ketamine treatments. Thirty healthy controls will also be studies at two points but will not receive treatment. Subjects will undergo a structural scan, resting state functional magnetic resonance imaging (fMRI) and Diffusion Weighted Imaging (DWI) scans at baseline and at the two time-points. In addition to imaging, using an innovative approach, we will also collect living neurons from olfactory epithelium using a soft nasal brushing procedure to conduct molecular and gene expression analysis. We will acquire imaging on a state-of-the-art 7-T scanner and apply cutting-edge brain network properties analyses and correlate with molecular changes as well as changes in depression scores. We will conduct a mediation analysis to identify specific molecular/gene expression alterations which cause connectome changes which in turn lead to rapid antidepressant and antisucidal effects. This study will therefore provide unique data regarding imaging and molecular correlates of rapid antidepressant action of ketamine. In addition, this mechanistic clinical trial will provide a new paradigm for treatment monitoring and drug development of novel rapidly acting antidepressant therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to give voluntary informed consent; 2. Satisfy criteria for Diagnostic and Statistical Manual 5th edition (DSM-V) for Major Depression Disorder (MDD) 3. Currently in a depressive episode (MDE); 4. Montgomery and Asberg Depression Rating Scale (MADRS) score >21 but <32(moderate to severe depression)11; 3. Psychotropic medication-free > 2weeks and if on fluoxetine then for >5 weeks at time of inclusion in the study(no taper or medication washout will be done for the purpose of the study). 6. Satisfy criteria to undergo an MRI scan based on MRI screening questionnaire; 7) able to be managed as outpatients during the study as ascertained by Clinical Global Severity Scale < 5 (i.e., moderately ill) and no suicidal/homicidal intent or behavior or gross disability; and 8) no contraindication to KET treatment such as KET allergy or uncontrolled hypertension.

Exclusion Criteria:

* 1. Meeting DSM-5 criteria for (hypo)mania, bipolar disorder, schizophrenia, schizophreniform disorder, schizoaffective disorder, intellectual disability, or pervasive developmental disorder; 2. History of receiving electroconvulsive therapy in the past 1 year (due to possible effects on brain morphology); 3. Meeting DSM-5 criteria for moderate or severe substance/alcohol use within the past 6 months excluding caffeine or nicotine. The criteria will be evaluated by interview and urinary toxicology screening. The typical weekly use of caffeine, nicotine and alcohol will be recorded; 4. No serious medical or neurological illness, including previously known HIV positive status (due to possible CNS involvement) as assessed by history, physical examination and laboratory examination including EKG, CBC and blood chemistry; 5. Current pregnancy or breast feeding; 6. Metallic implants or contraindication to MRI.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Rating Scale (MADRS) | From enrollment to end of 1 week treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hosipital, Boston, Massachusetts, United States